CLINICAL TRIAL: NCT02057666
Title: A Phase III, Randomised, Double-Blind, Placebo-Controlled Study Of Tasquinimod In Asian Chemo-Naïve Patients With Metastatic Castrate-Resistant Prostate Cancer
Brief Title: Study Of Tasquinimod In Asian Chemo-Naïve Patients With Metastatic Castrate-Resistant Prostate Cancer
Acronym: TasQ003
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Development of tasquinimod in prostate cancer discontinued
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8-55-58102-003
Record Dates: First submitted 2014-02-06; First posted 2014-02-07 (Estimated); Results first posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-03

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: CRPC; Metastatic; Chemotherapy naïve; Chemo-naïve; Prostate cancer; mCRPC; Chemotherapy-naïve; Chemo naïve
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Neoplasm Metastasis; Prostatic Neoplasms | interventions — tasquinimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tasquinimod (Experimental): One capsule (0.25, 0.50 or 1 mg), taken orally once a day with water and food (preferably the main evening meal).
  Interventions: Drug: Tasquinimod
- Placebo (Placebo Comparator): One capsule, taken orally once a day with water and food (preferably the main evening meal).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tasquinimod — A patient initially received a 0.25 mg/day dose which was then titrated through 0.5 mg/day (from Day 15) to a maximum of 1 mg/day (from Day 29). If tolerability issues arose at 0.5 or 1 mg/day, patients had their dose reduced to 0.25 or 0.5 mg/day, respectively.
  Other Names: ABR-215050
  Arms: Tasquinimod
Drug: Placebo — Placebo capsules were identical to tasquinimod capsules in appearance and excipients but excluded the active compound (tasquinimod).
  Arms: Placebo

SUMMARY:
The primary objective was to confirm the effect of tasquinimod in delaying disease progression or death as compared with placebo in chemo-naïve patients with metastatic castrate-resistant prostate cancer (mCRPC).

Secondary objectives included further evaluation of the safety profile of tasquinimod, comparison of clinical benefits (such as overall survival and symptoms) of tasquinimod with placebo, to evaluate the quality of life impact and to determine the pharmacokinetics of tasquinimod.

DETAILED DESCRIPTION:
The study involved a 4-week Screening Period, Baseline Visit (Day 1) where the patient was randomised, followed by a Double Blind Treatment Period. Patients initially received tasquinimod (or corresponding placebo) at a 0.25 mg/day dose which was then titrated through 0.5 mg/day (from Day 15) to a maximum of 1 mg/day (from Day 29). If tolerability issues arose at 0.5 or 1 mg/day, patients had their dose reduced to 0.25 or 0.5 mg/day, respectively. The Double Blind Treatment Period continued until the death of the patient or any criterion for withdrawal from study treatment was reached. Any placebo treated patients with radiological disease progression confirmed by the central imaging assessment, who remained asymptomatic or mildly symptomatic were, at the Investigator's discretion, given the option to continue on active treatment (tasquinimod) during an Open-Label Treatment Period, following the same titration rule described above until progression under active treatment. All other patients stopped study treatment.

An End-of-Study Treatment/Withdrawal Visit was to be performed within 14 days after the last dose of study treatment and patients were then to be followed up every 6 months until 80% of the patients had died or 2 years after the last patient was randomised, whichever occurred last.

A PK ancillary study was to be performed in a subgroup of 12 Asian-Chinese patients before randomisation; however, due to the early termination of this study, only some samples were analysed and no PK analyses were performed.

ELIGIBILITY:
Inclusion Criteria:

1. Asian male aged at least 20 years at the time of signing the informed consent form.
2. Histologically confirmed diagnosis of adenocarcinoma of the prostate.
3. Evidence of metastatic disease (bone and/or visceral), excluding node lesion only, on radiographic examination, whether from bone scan (bone lesions) or other imaging modality (CT scan/MRI).
4. Chemical or surgical castration verified by levels of serum testosterone ≤50 ng/dL (1.75 nmol/L).
5. Evidence of progressive disease after castration levels of testosterone had been achieved, defined by any of the following criteria:

   * Increasing serum Prostate Specific Antigen (PSA) levels, with the most recent value ≥2 ng/mL (increasing levels must have been confirmed by three consecutive PSA measurements, within 15 months prior to the start of study treatment. The time between each PSA test should have been preferably at least 14 days, however a minimum of 7 days was acceptable. The third value was used for study selection).
   * Progression of soft tissue metastasis documented within 6 weeks prior to randomisation (CT scan or MRI).
   * Progression of bone disease (at least one new bone lesion as measured by bone scan within the 12 weeks prior to the start of study treatment).
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Laboratory values as follows:

   * Haemoglobin ≥90 g/L (≥9 g/dL).
   * Absolute neutrophil count ≥1500/μL.
   * Platelets ≥100,000/μL.
   * Serum creatinine ≤1.5 times the upper limit of normal (ULN).
   * Total bilirubin ≤1.5 times ULN.
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 times ULN (≤5 times ULN if liver metastases were present).
   * Serum amylase ≤ULN (if serum amylase >ULN, pancreatic amylase and serum lipase should have been analysed. If both pancreatic amylase and serum lipase were >ULN, patient excluded).
8. If sexually active with partner of childbearing potential, patient agreed to use adequate contraceptive method (barrier contraceptive with spermicide) while receiving study treatment and until 14 days after the stop of study treatment or had been previously vasectomised.
9. No evidence (within last 5 years) of prior malignancies (except successfully treated basal cell or squamous cell carcinoma of the skin).
10. Able to swallow and retain oral medication.
11. Able to adhere to the study visit schedule and other protocol requirements.
12. Ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to cooperate with the Investigator and to comply with the requirements of the entire study.
13. Able to sign and date the written informed consent after being informed of the full nature and purpose of the study, including possible risks and side effects, and given ample time and opportunity to read and understand this information.

Exclusion Criteria:

1. Cytotoxic chemotherapy for the treatment of prostate cancer within 2 years prior to the start of study treatment.
2. Previous anticancer therapy using radiation, biologics or vaccines and including sipuleucel-T (Provenge®) within 4 weeks prior to the start of study treatment and abiraterone, TAK700 or MDV3100 within 2 weeks prior to the start of study treatment. Before inclusion, abiraterone, TAK700 or MDV3100 related adverse effect must have been resolved to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 Grade ≤1. If radiation therapy was applied after Baseline scan, a new Baseline scan needed to be done at least 4 weeks after the radiation therapy.
3. Therapy with antiandrogens within 4 weeks (within 6 weeks for bicalutamide e.g. Casodex®) prior to the start of study treatment.
4. Concurrent use of other anticancer agents or treatments, with the exception of ongoing treatment with luteinising hormone-releasing hormone (LHRH) agonists or antagonists, denosumab (Prolia®) or bisphosphonate (e.g. zoledronic acid), which were allowed. Ongoing treatment was to be kept at a stable schedule; however, if medically required, a change of dose, compound, or both was allowed.
5. Any treatment modalities involving major surgery within 4 weeks prior to the start of study treatment.
6. Prostate cancer pain that required ongoing treatment with narcotic analgesics or warranted the initiation of radio- or chemotherapy.
7. Both of the following criteria:

   * Visceral metastasis.
   * Bone lesions both on and outside of the spinal axis.
8. PSA >100 ng/mL.
9. Ongoing treatment with warfarin.
10. Maintenance treatment with corticosteroids corresponding to a prednisolone or prednisone dose above 10 mg/day. The dose must have been stable for at least 5 days.
11. Systemic exposure to ketoconazole or other strong cytochrome P450 (CYP) 3A4 isozyme inhibitors or inducers within 14 days prior to the start of study treatment. Systemic exposure to amiodarone was not allowed within 1 year prior to the start of study treatment.
12. Ongoing treatment with sensitive CYP1A2 substrate or CYP1A2 substrate with narrow therapeutic range at the start of study treatment.
13. Ongoing treatment with CYP3A4 substrate with narrow therapeutic range at the start of study treatment.
14. Simultaneous participation in any other study involving treatment with investigational drugs or having received treatment with investigational drugs less than 4 weeks prior to the start of study treatment.
15. Myocardial infarction, percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass graft, New York Heart Association (NYHA) class III/IV congestive heart failure, cerebrovascular accident, transient ischaemic attack, or limb claudication at rest, within 6 months prior to start of study treatment, history of venous thrombo-embolic disease within 3 months prior to randomisation and ongoing symptomatic dysrhythmias, unstable angina, uncontrolled hypertension, and uncontrolled atrial or ventricular arrhythmias.
16. History of pancreatitis.
17. Known brain or epidural metastases.
18. Known positive serology for human immunodeficiency virus (HIV) (patients with known history of HIV were excluded because of potential for unforeseen toxicity and morbidity in an immunocompromised host).
19. Chronic hepatitis with advanced, decompensated hepatic disease or cirrhosis of the liver or history of a chronic viral hepatitis or known viral hepatitis carrier (patients who had recovered from hepatitis were allowed to enter the study) with abnormal liver function.
20. Patients with active tuberculosis (TB), or with known, untreated latent TB (country-specific TB therapy should have been given for at least 30 days prior to the start of study treatment and the patient should have intended to complete the entire course of that therapy).
21. Any condition, including other active or latent infections, medical or psychiatric conditions, or the presence of laboratory abnormalities, which could have confounded the ability to interpret data from the study or placed the patient at unacceptable risk if he participated in the study.
22. Any patient who in the opinion of the Investigator should not have participated in the study.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Uro-Oncology, Study Director — Ipsen
Locations (36):
- China (27):
  - Beijing Chao-Yang Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Hospital of Ministry of Health, Beijing, Beijing Municipality
  - Southwest Hospital (the First Affiliated Hospital of Third Military Medical University PLA), Chongqing, Chongqing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangshou First People's Hospital, Guangzhou, Guangdong
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Ruijin Hospital Shanghai Jiaotong University of Medicine, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Huadong Hospital Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Sichuan Academy of Sichuan Medical Sciences & Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - General Hospital Chengdu Military Region of PLA, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital College of Medicine Zhujiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- South Korea (5):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheong Province
  - Chonnam National University Hospital, Gwangju
  - Gangnam Severance Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited across 36 centres. The first patient first visit was on 24 January 2014. The last patient was randomised into the study on 16 April 2015; however, early termination of the study was announced on the same day. Due to a necessary visit for 1 patient, the last patient last visit of the study was on 26 May 2015.
Pre-assignment Details: 229 patients were screened, of whom 146 were randomised (96 tasquinimod, 50 placebo).
Groups:
- Tasquinimod: One capsule (0.25, 0.50 or 1 mg), taken orally once a day with water and food (preferably the main evening meal).
  A patient initially received 0.25 mg/day dose which was then titrated through 0.5 mg/day (from Day 15) to a maximum of 1 mg/day (from Day 29). If tolerability issues arose at 0.5 or 1 mg/day, patients had their dose reduced to 0.25 or 0.5 mg/day, respectively.
Period: Double Blind Treatment Period
Arm/Group | Tasquinimod | Placebo
Started | 96 | 50
Completed | 0 (Number of patients who continued into the open-label treatment period.) | 6 (Number of patients who continued into the open-label treatment period.)
Not Completed | 96 | 44
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Poor tolerability | 7 | 2
Not completed — Symptomatic disease progression | 8 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Progressive disease for bone lesion | 1 | 0
Not completed — Subject planning to withdraw | 1 | 0
Not completed — Sponsor's request | 70 | 34
Period: Open-Label Treatment Period
Arm/Group | Tasquinimod | Placebo
Started | 0 | 6
Completed | 0 | 0
Not Completed | 0 | 6
Not completed — Poor tolerability | 0 | 1
Not completed — Symptomatic disease progression | 0 | 1
Not completed — Sponsor's request | 0 | 4

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population: All randomised patients. Patients were allocated to the treatment they were randomised to. This population consisted of all randomised patients regardless of whether or not the patient received any dose of the study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tasquinimod | Placebo | Total
Number analyzed (Participants) | 96 | 50 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 9 | 25
  >=65 years | 80 | 41 | 121
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 96 | 50 | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 96 | 50 | 146
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 69 | 34 | 103
  Taiwan | 5 | 5 | 10
  Korea, Republic of | 22 | 11 | 33
Status of Visceral Metastases [Count of Participants; unit: Participants] — Evidence of metastatic disease on radiographic examination, whether from bone scan (bone lesions) or other imaging modality (computed tomography [CT] scan/magnetic resonance imaging [MRI]).
  Participants
    Presence | 4 | 2 | 6
    Absence | 92 | 48 | 140

OUTCOME MEASURES:

1. Primary Outcome: Time to Radiological Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of randomisation to the date of radiological progression (confirmed by the central imaging assessment) or death due to any cause. Radiological progression was defined by any of the following criteria: progression of soft tissue lesions evaluated by computed tomography (CT) or magnetic resonance imaging (MRI) scan according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 criteria; progression of bone lesions detected with bone scan according to Prostate Cancer Clinical Trials Working Group 2 (PCWG2) criteria; or radiologically confirmed spinal cord compression or pathological fracture due to malignant progression.
  The primary endpoint was centrally and independently evaluated.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
Population: ITT population: All randomised patients. Patients were allocated to the treatment they were randomised to. This population consisted of all randomised patients regardless of whether or not the patient received any dose of the study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tasquinimod | Placebo
Number analyzed (Participants) | 96 | 50
months | 11.00 [11.00 to NA] — The upper 95% confidence interval limit could not be calculated due to too few participants with events. | 7.53 [5.67 to NA] — The upper 95% confidence interval limit could not be calculated due to too few participants with events.
Statistical Analysis 1: Comparison: Tasquinimod vs Placebo; Test type: Superiority or Other; p = 0.027, Log Rank; Stratified as per randomisation; Hazard Ratio (HR) = 0.406, 95% CI 2-sided [0.182 to 0.903] — Stratified as per randomisation

2. Secondary Outcome: Overall Survival
Description: An overall survival event was defined as death due to any cause. The number of participants with overall survival events is reported.
Time Frame: From randomisation up to 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tasquinimod | Placebo
Number analyzed (Participants) | 96 | 50
Participants
  Number of deaths | 2 | 2
  Number of censored observations | 94 | 48
Statistical Analysis 1: Comparison: Tasquinimod vs Placebo; Test type: Superiority or Other; p = 0.448, Log Rank; Hazard Ratio (HR) = 0.465, 95% CI 2-sided [0.065 to 3.355]

3. Secondary Outcome: Local Assessment of Radiological PFS
Description: The Investigator was to evaluate radiological disease progression in accordance with the criteria defined for the primary endpoint.
Time Frame: as for outcome 1
Population: No data collected due to the early termination of the study. Therefore, no analyses performed on this secondary efficacy endpoint.
Arm/Group | Tasquinimod | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Symptomatic PFS Based on Local Assessment
Description: Symptomatic PFS, defined as the time from the date of randomisation to the date of appearance of pain (using pain visual analogue scale (VAS)) at a site with documented disease and analgesic use, or skeletal-related events, or death due to prostate cancer, whichever occurred first.
Time Frame: Every 3 months
Population: as for outcome 3
Arm/Group | Tasquinimod | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time From Randomisation to Further Treatment for Prostate Cancer
Description: The need for any anti-tumour prostate cancer treatments was to be recorded during the Follow-up Period, with the time to further treatment to subsequently be derived.
Time Frame: Every 6 months during the follow-up period
Population: as for outcome 3
Arm/Group | Tasquinimod | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Quality of Life (QoL)
Description: QoL measured by the Functional Assessment of Cancer Therapy Prostate Module (FACT-P) questionnaire and by the EuroQol 5-Dimension QoL Instrument (EQ-5D).
  Due to the early termination of the study, a simplified data analysis (primary endpoint and overall survival) was performed to fulfil the requirement from regulatory authorities for early termination studies. Therefore, no analyses were performed on this secondary efficacy endpoint.
Time Frame: Every 3 months
Reporting Status: Not Posted

7. Secondary Outcome: Tasquinimod Pharmacokinetic (PK) Profile
Description: Tasquinimod PK profile:
  1. Following a single 1 mg dose of tasquinimod given to a subgroup of 12 Asian-Chinese patients (ancillary study).
  2. At steady state conditions based on limited sampling strategy.
  Following termination of the study the PK analyses were not performed.
Time Frame: Up to 216 hours after a single dose and during the double blind treatment period (Day 15, 29, 57 and 127)
Population: as for outcome 3
Arm/Group | Tasquinimod | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were monitored from informed consent until the date of death from any cause or 14 days after the last dose of study treatment, whichever came first, assessed up to 2 years.
Description: AEs were elicited by direct, non-leading questioning or by spontaneous reports. Natural progression/deterioration of the malignancy and death due to disease progression were to be recorded as part of the efficacy evaluation (not an AE/serious AE (SAE)).
  Non-serious AEs were not available. Therefore all TEAEs are presented Adverse Events section.
  Safety analyses were provided for the Double-Blind Period. Due to early termination, only 6 patients entered the Open-Label Period.
Arm/Group | Tasquinimod | Placebo
All-Cause Mortality (participants affected / at risk) | 76/94 | 30/50
Serious Adverse Events (participants affected / at risk) | 19/94 | 5/50
Other Adverse Events (participants affected / at risk) | 52/94 | 19/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tasquinimod (N=94) | Placebo (N=50)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Radiculitis (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tasquinimod (N=94) | Placebo (N=50)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 6 (7) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (7) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 3 (4)
Asthenia (General disorders) | 5 (5) | 1 (2)
Oedema peripheral (General disorders) | 5 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 2 (5)
Haemoglobin decreased (Investigations) | 1 (1) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 16 (18) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (17) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (12) | 1 (1)
Pain in extemity (Musculoskeletal and connective tissue disorders) | 6 (8) | 5 (5)
Dysuria (Renal and urinary disorders) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
The study was terminated early due to the Sponsor deciding to stop development in prostate cancer; therefore, the results of all efficacy analyses should be considered exploratory and not supportive of efficacy in any indication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor required reasonable opportunity to review any abstract, presentation, or paper before the material was submitted for publication or communicated. This also applied to any amendments that were requested by referees or journal editors. The Sponsor committed to comment on the draft documents within a time period agreed in the contractual arrangements between the Sponsor and authors or their institution. Delays were also possible if publication would adversely affect patentability.